CLINICAL TRIAL: NCT03947268
Title: Palliative Short-course Radiotherapy in Advanced Pelvic Cancer: a Phase II Study (SHARON Project)
Brief Title: Radiotherapy in Palliation of Advanced Pelvic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARON PELVIS (phase II trial)
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Palliative Care
Keywords: palliative care; pelvic cancer; radiotherapy; pain; Quality of life
MeSH Terms: conditions — Pelvic Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-course radiotherapy (Experimental): The radiotherapy is delivered over 2 days with accelerated hypo-fractionation technique.
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — An accelerated hypo-fractionation 2D-radiotherapy is delivered for palliation in patients with advanced pelvic cancer.

SUMMARY:
The study wants to define the safety and efficacy of a short-course radiation therapy in patients with symptomatic advanced pelvic cancer.

DETAILED DESCRIPTION:
he study wants to define the safety and efficacy of a short course accelerated radiation therapy delivered in twice daily fractions and 2 consecutive days for symptomatic palliation of advanced solid cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven advanced pelvic cancer
* excluded from curative therapy because of disease stage and/or presence of multiple comorbidities and/or poor performance status
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) <3

Exclusion Criteria:

- prior radiotherapy to the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of symptoms [pain] | 1 year]
  Pain after treatment is evaluated with the Visual Analogic scale (VAS). Values range from 0 (no pain) to 10 (maximum possible pain).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Acute radiation toxicity] | 1 year
  Acute toxicity after treatment is evaluated with the Common Terminology Criteria for Adverse Events (CTCAE). Values range from 1 (minimum acute toxicity) to 5 (maximum acute toxicity).
Incidence of Treatment-Emergent Adverse Events [Late radiation toxicity] | 1 year
  Late toxicity after the treatment is evaluated with the Toxicity criteria of the Radiation Therapy Oncology Group and the European Organization for Research and Treatment of Cancer (RTOG/EORTC). Values range from 1 (minimum late toxicity) to 5 (maximum/severe late toxicity).
Assessment of the Quality of life (QOL) | 1 year
  Quality of life after the treatment is evaluated according with the Cancer Linear Analog Scale (CLAS). CLAS scale evaluates well-being, fatigue, and ability to perform daily activities. This method is based on a linear analogue scale. Values range from 0 (better status) to 10 (worst status).

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, S.Orsola-Malpighi Hospital, Bologna, Italy